CLINICAL TRIAL: NCT00177307
Title: Phase II Study of the A-ICOX Regimen Consisting of Bevacizumab (Avastinâ), Intermittent Dose Capecitabine (Xelodaâ) and Oxaliplatin (Eloxatinâ) in Patients With Untreated Advanced Colorectal Cancer
Brief Title: Safety and Efficacy Study Using Bevacizumab, Capecitabine and Oxaliplatin for Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Nathan Bahary, MD, Associate Professor, Department of Medicine, Division of Oncology, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-118
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Cancer
Keywords: colon; rectum
MeSH Terms: conditions — Neoplasms | interventions — Bevacizumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxaliplatin, Capecitabine, and Bevacizumab (Experimental)
  Interventions: Drug: Bevacizumab; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 5 mg/kg by 90-30 minute IV infusion IV q 2 weekly Until disease progression or unacceptable toxicity
  Other Names: Capecitabine 2500 mg/m2/d in two divided doses; (May be 2000 or 3000 mg/m2/d after interim analysis) Days 1-8, every 2 weeks Until disease progression or unacceptable toxicity; Oxaliplatin 85 mg/m2 IV q 2 weekly Until disease progression, unacceptable toxicity,; or Grade 3 neuropathy or cumulative dose of 1200 mg/m2
Drug: Capecitabine — Capecitabine will be administered orally at twice daily 1250 mg/m2 (equivalent to a total daily dose of 2500 mg/m2) as intermittent therapy (1 week of treatment followed by one week without treatment) and this cycle repeated every 14 days. The first dose of capecitabine will be given on day 1 of each cycle as evening dose and the last dose will be given on day 8 as morning dose (for a total of 14 single doses per cycle).
Drug: Oxaliplatin — Oxaliplatin will be administered at the dose of 85 mg/m2 given as a 2-hour intravenous infusion on day 1 of a two-week cycle, prior to the first dose of capecitabine

SUMMARY:
This is a Phase II study of the drug combination of Oxaliplatin, Avastin and capecitabine. This is an open-label study.

DETAILED DESCRIPTION:
Ongoing clinical trials are now evaluating the addition of bevacizumab to standard chemotherapeutic regimens for colorectal cancer such as FOLFOX or FOLFIRI. In these studies the addition of bevacizumab has been safe and has not resulted in significantly increased toxicity. Our proposed regimen has the advantage of being easily administered in the outpatient setting, with potential for enhanced activity and needs to be evaluated in a clinical trial.

The patterns of care for CRC have shifted, IFL previously the standard of care, is now proven to be an inferior regimen compared to FOLFOX4. (8) The recent FDA approval in February 2004 of bevacizumab for first line therapy, which states that bevacizumab is an approved agent in combination with a 5-FU regimen, gives no clear guidelines as to the "best regimen". This is an issue that needs to be evaluated rapidly in clinical trials, and it is clear that a combination of 5-FU or capecitabine with oxaliplatin and bevacizumab is one of the most active and well-tolerated regimens. The optimum sequence, schedule and doses needs to determined in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* advanced, surgically unresectable CRC
* measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension(histological confirmation of adenocarcinoma of the colon or rectum.

ECOG performance status of 0, 1, or 2 Estimated life expectancy of at least 12 weeks.

* chemotherapy prior to the diagnosis of metastatic disease. The chemotherapy regimen must not have included oxaliplatin or bevacizumab. No prior therapy for metastatic disease is permitted.
* Evidence of adequate organ function, including:
* Evidence of adequate hepatic function,
* Evidence of adequate renal function INR <1.5 x ULN (unless taking warfarin in which case it must be in the therapeutic range). Patients on warfarin are allowed to participate.
* Absence of proteinuria on urine analysis· Patients with a history of prior non-colorectal malignancies are eligible if they have been disease-free for at least 5 years prior to study entry and are deemed by the physician to be at low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: melanoma in situ, and basal cell and squamous cell carcinoma of the skin.
* Age > 18 yrs.

Exclusion Criteria:

* Any systemic therapy administered for metastatic or locally recurrent disease. Patients who are considered candidates for surgical resection of metastatic and/or locally advanced disease.
* Any histology other than adenocarcinoma of the colon or rectum.
* Pregnancy or lactation at the time of patient entry or women of childbearing potential with no pregnancy test. Eligible patients of reproductive potential (both sexes) must agree to use adequate contraceptive methods during and for 6 months after study therapy.
* Serious concomitant medical conditions that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study.
* General Medical Concerns History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.
* Serious, uncontrolled, concurrent infection.
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study; fine needle aspirations or core biopsies within 7 days prior to Day 0.
* Proteinuria at baseline or clinically significant impairment of renal function.
* Serious, non healing wound, ulcer, or bone fracture
* Subjects who can not take oral medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Bahary, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 40 patients were enrolled, but one subject withdrew before starting therapy.
Period: Overall Study
Arm/Group | Oxaliplatin, Capecitabine, and Bevacizumab
Started | 40
Completed | 39
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oxaliplatin, Capecitabine, and Bevacizumab
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 62 [38 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: time from start of protocol therapy until objective tumor progression or death
Time Frame: Up to 27 Months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Oxaliplatin, Capecitabine, and Bevacizumab
Number analyzed (Participants) | 39
Months | 8.6 [4.7 to 10.2]

2. Secondary Outcome: Response Rate (RR)
Description: Percentage of partial responses (PR) + complete responses (CR).
Time Frame: Up to 27 months
Measure: Number; unit: percentage of participants
Arm/Group | Oxaliplatin, Capecitabine, and Bevacizumab
Number analyzed (Participants) | 39
percentage of participants | 38

3. Secondary Outcome: Overall Survival
Description: time from start of protocol therapy until death from any cause
Time Frame: Up to 40 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Oxaliplatin, Capecitabine, and Bevacizumab
Number analyzed (Participants) | 39
Months | 17.2 [10.4 to 24.2]

4. Secondary Outcome: 1-, 2-, and 3-year Overall Survival
Description: Probability of being alive at 1-, 2-, and 3-years from start of protocol therapy
Time Frame: Up to 40 months
Measure: Number; unit: percent chance
Arm/Group | Oxaliplatin, Capecitabine, and Bevacizumab
Number analyzed (Participants) | 39
percent chance
  1 year-overall survival | 62
  2 year-overall survival | 36
  3 year-overall survival | 24

ADVERSE EVENTS:
Arm/Group | Oxaliplatin, Capecitabine, and Bevacizumab
Serious Adverse Events (participants affected / at risk) | 25/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin, Capecitabine, and Bevacizumab (N=39)
Anemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Investigations) | 2
Diarrhea (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 4
Neuropathy (Nervous system disorders) | 4
Bowel perforation (Gastrointestinal disorders) | 1
Bleeding (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin, Capecitabine, and Bevacizumab (N=39)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1
Alkaline phosphatase (Investigations) | 1
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2
Amylase (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 18
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 2
Ataxia (incoordination) (Nervous system disorders) | 1
Auditory/Ear - Other (Ear and labyrinth disorders) | 1
Bilirubin (hyperbilirubinemia) (Investigations) | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1
Coagulation - Other (Blood and lymphatic system disorders) | 2
Constipation (Gastrointestinal disorders) | 11
Constitutional Symptoms - Other (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Cystitis (Renal and urinary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 2
Diarrhea (Gastrointestinal disorders) | 16
Dizziness (Nervous system disorders) | 8
Dry eye syndrome (Eye disorders) | 1
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4
Edema: limb (General disorders) | 3
Fatigue (asthenia, lethargy, malaise) (General disorders) | 27
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10^9 cells/L) (General disorders) | 8
Flatulence (Gastrointestinal disorders) | 2
Flushing (Vascular disorders) | 1
Gastrointestinal - Other (Gastrointestinal disorders) | 2
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 8
Hemoglobin (Blood and lymphatic system disorders) | 14
Hemorrhage, GI, Lower GI NOS (Gastrointestinal disorders) | 1
Hemorrhage, pulmonary/upper respiratory, Mediastinum (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, pulmonary/upper respiratory, Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage/Bleeding - Other (Blood and lymphatic system disorders) | 1
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Blood (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Joint (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Lung (pneumonia) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Oral cavity-gums (gingivitis) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Sinus (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Skin (cellulitis) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Upper airway NOS (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Urinary tract NOS (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Wound (Infections and infestations) | 1
Injection site reaction/extravasation changes (General disorders) | 7
Joint-effusion (Musculoskeletal and connective tissue disorders) | 1
Leukocytes (total WBC) (Investigations) | 12
Lipase (Investigations) | 1
Mood alteration, Anxiety (Psychiatric disorders) | 3
Mood alteration, Depression (Psychiatric disorders) | 3
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 2
Muscle weakness, generalized or specific area (not due to neuropathy), Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 22
Neurology - Other (Nervous system disorders) | 14
Neuropathy: motor (Nervous system disorders) | 2
Neuropathy: sensory (Nervous system disorders) | 23
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 11
Obstruction, GI, Small bowel NOS (Gastrointestinal disorders) | 1
Ocular/Visual - Other (Eye disorders) | 3
Pain - Other (General disorders) | 2
Pain, Abdomen NOS (Gastrointestinal disorders) | 12
Pain, Back (Musculoskeletal and connective tissue disorders) | 3
Pain, Bone (Musculoskeletal and connective tissue disorders) | 2
Pain, Buttock (Musculoskeletal and connective tissue disorders) | 1
Pain, Chest/thorax NOS (General disorders) | 1
Pain, Extremity-limb (Musculoskeletal and connective tissue disorders) | 5
Pain, Face (General disorders) | 1
Pain, Head/headache (Nervous system disorders) | 2
Pain, Joint (Musculoskeletal and connective tissue disorders) | 1
Pain, Muscle (Musculoskeletal and connective tissue disorders) | 2
Pain, Neck (Musculoskeletal and connective tissue disorders) | 1
Perforation, GI, Small bowel NOS (Gastrointestinal disorders) | 0
Platelets (Investigations) | 7
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 16
Renal/Genitourinary - Other (Renal and urinary disorders) | 3
Rigors/chills (General disorders) | 5
Seizure (Nervous system disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2
Somnolence/depressed level of consciousness (Nervous system disorders) | 1
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1
Supraventricular and nodal arrhythmia, Atrial tachycardia/Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 2
Syncope (fainting) (Nervous system disorders) | 1
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 6
Tremor (Nervous system disorders) | 2
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 16
Weight gain (Investigations) | 1
Weight loss (Investigations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes